CLINICAL TRIAL: NCT02308345
Title: MiVideo - Video Visit Summary for Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Lawrence C. An, Director, Center for Health Communications Research, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00090259
Record Dates: First submitted 2014-10-22; First posted 2014-12-04 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video summary (Experimental): Participants in this arm will be given online access to a 5-minute video summary of their pre-chemotherapy visit, recorded by their physician.
  Interventions: Other: Pre-chemotherapy visit summary Video

INTERVENTIONS:
Other: Pre-chemotherapy visit summary Video

SUMMARY:
Cancer patients about to begin chemotherapy receive large amounts of information regarding their prognosis, how chemotherapy improves their prognosis, and the usual side effects of the chemotherapy during their first visit to the oncologist. Prior studies have documented that less than half of this information is retained after the visit, making it difficult for patients to participate in their care and difficult for them to enlist the help of their social support. The MiVideo project allows the physician to create a custom 5-minute summary video summary of a pre-chemotherapy clinic visit and upload it to a secure web site. The video will emphasize the major points of the forty-five minute office discussion, allowing patients to review the physicians' recommendations and share the information and recommendations with others. By providing the patient with this re-cap of their visit, the investigators hope to engage them more actively in their cancer treatment. Making the information available to friends and family can also help a patient receive both intellectual and emotional support during the course of treatment. The primary endpoint of this study is improvement of patient care, not research activity.

Primary Hypothesis: Creating a 5-minute video summarizing information about diagnosis, stage, chemotherapy treatment plan, and anticipated side effects for patients starting chemotherapy for colon cancer will not significantly lengthen the pre-chemotherapy clinic visit as compared to visits that do not include video production.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Diagnosis of colon cancer with treatment plan to include chemotherapy
* Sufficient command of English language to read and understand consent and survey forms
* Working email address and access to the Internet (computer, tablet, smartphone) to view treatment summary video

Exclusion Criteria:

* Previous history of chemotherapy or cancer (excepting in situ cancers)
* History of drug or alcohol abuse or unmedicated mental or psychiatric disorder
* Medical history or diagnosis of debilitating medical disorder such as progressive muscle paralysis, advanced cardiac, respiratory, or renal disease, or AIDS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Length of visit (minutes) | Day of consent

SECONDARY OUTCOMES:
Number of patient views of their visit summary prior to chemotherapy | 2-4 weeks post-visit
Number of video summary shares prior to chemotherapy | 2-4 weeks post visit
Participant-rated usefulness of video summary | 2-4 weeks post visit
  Usefulness is measured using a short post-video online survey.

CONTACTS AND LOCATIONS:
Overall Officials: Larry C An, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided